CLINICAL TRIAL: NCT06298123
Title: Risk Factor Analysis and Prognostic Modelling of Postoperative Adjuvant Immunotherapy for Hepatocellular Carcinoma
Brief Title: Postoperative Adjuvant Immunotherapy for Hepatocellular Carcinoma: Risk Factor Analysis and Prognostic Modelling
Status: Completed | Type: Observational
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: adjuvant-03
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma; Adjuvant Immunotherapy; Checkpoint Inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — spartalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anti-PD-1 monoclonal antibody — The independent risk factors for hepatocellular carcinoma (HCC) patients undergoing adjuvant immunotherapy after hepatic resection surgery were analysed by retrospectively collecting patient data from the Centre for Liver Surgery, Tongji Hospital, during the period of February 2019 to February 2023, and comprehensively evaluating the patients' demographic characteristics, oncological parameters, surgical details, and response to immunotherapy, and establishing a prognostic model based on these factors.
  Other Names: Prognostic analysis

SUMMARY:
The aim of this study was to analyse the independent risk factors for hepatocellular carcinoma (HCC) patients undergoing adjuvant immunotherapy after liver resection surgery, and to develop a prognostic model based on these factors.

DETAILED DESCRIPTION:
By retrospectively collecting patient data from a single centre of liver surgery at Tongji Hospital between February 2019 and February 2023, the study aimed to comprehensively evaluate patients' demographic characteristics, oncological parameters, surgical details and response to immunotherapy to identify the key factors affecting postoperative recurrence and survival.

ELIGIBILITY:
Inclusion Criteria:

* HCC confirmed by pathologists
* Undergone a curative resection (R0)
* Aged 18-75 years
* No previous systematic treatment and locoregional therapy for HCC prior to randomization
* Absence of major macrovascular invasion
* No extrahepatic spread

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, mixed cholangiocarcinoma or recurrent HCC
* Any preoperative treatment for HCC including local and systemic therapy
* Unable to receive adjuvant therapy due to surgery-related complications, acute active infectious diseases, active or history of autoimmune disease, or immune deficiency
* incomplete clinical data

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma (HCC) who underwent radical hepatectomy with adjuvant immunotherapy at the Liver Surgery Centre of Tongji Hospital between February 2019 and February 2023.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | 2019-2023
  RFS is defined as the time from randomization to the first documented occurrence of local, regional, or metastatic HCC as determined by BIRC, or death from any cause (whichever occurs first).

SECONDARY OUTCOMES:
Overall Survival (OS) | 2019-2023
  OS is defined as the time from randomization to death from any cause

OTHER OUTCOMES:
Imaging data (enhanced CT and MRI） and histopathology data, if available. | 2019-2023
  Pre-surgical imaging data will be collected for machine learning to synthesise imaging features prognostic factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China